CLINICAL TRIAL: NCT04267146
Title: Phase I-II Study of Nivolumab in Combination With Temozolomide and Radiotherapy in Children and Adolescents With Newly Diagnosed High-grade Glioma
Brief Title: Nivolumab in Combination With Temozolomide and Radiotherapy in Children and Adolescents With Newly Diagnosed High-grade Glioma
Acronym: NIVOGLIO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002688-24; 2019/2797 (Other: CSET number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — Nivolumab; Temozolomide; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Multicenter, open label, prospective study including successively a phase I trial and then a phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- newly diagnosed high-grade glioma (Experimental): Phase I : Open label, non-randomized, safety run study in nine patients. In case of safety issue a -1 dose level will be tested.
  Phase II : Open label, non randomized, efficacy study of nivolumab in addition to radiotherapy and temozolomide. This phase will start when the RP2D has been defined after the last patients evaluable for DLT achieved the first 6 weeks of treatment (the radio-chemotherapy period) with a DLT rate below 30% during the the phase I study.
  Interventions: Drug: Nivolumab; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nivolumab — Solution for intravenous injection 10 mg/ml. Initial dose : 3 mg/kg Nivolumab will be given at 3 mg/kg/injection every two weeks from the first day of radiotherapy to the last day of chemotherapy.
  One de-escalation dose : 1 mg/kg
Drug: Temozolomide — Capsules: 5, 20, 100, 140, 180 and 250 mg orally. Temozolomide will be given at 75mg/m2/day from the day of start of radiotherapy to the last day of radiotherapy, then, after one month rest at 200mg/m2/day for five consecutive days for 12 cycles (28 days cycle).
Radiation: Radiotherapy — Total dose of 54 Gray(Gy) units delivered in 30 daily fractions of 1.8 Gy over 6 weeks during the chemoradiation period.

SUMMARY:
Multicenter, open label, prospective study including successively a phase I trial and then a phase II trial Phase I : Open label, non-randomized, safety run study in nine patients. In case of safety issue a -1 dose level will be tested.

Phase II : Open label, non randomized, efficacy study of nivolumab in addition to radiotherapy and temozolomide. This phase will start when the RP2D has been defined after the last patients evaluable for DLT achieved the first 6 weeks of treatment (the radio-chemotherapy period) with a DLT rate below 30% during the the phase I study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific screening procedures are conducted according to local, regional or national guidelines
2. Age at inclusion: >/= 3 to <18 years of age
3. Patients should be able and willing to comply with study visits and procedures as per protocol.
4. Patients must be affiliated to a social security system or beneficiary of the same according to local requirements
5. Sexually active females of childbearing potential must have a negative serum pregnancy test within 24 hours prior to initiation of treatment. Sexually active women of childbearing potential must agree to use acceptable and appropriate contraception during the study and for at least 5 months after the last study treatment administration. Sexually active males patients (and their female partner) must agree to use condom during the study and for at least 7 months after the last study treatment administration.
6. Newly diagnosed non-brainstem WHO grade III and IV HGG and neuroglial tumors; gliomatosis cerebri or diffuse glioma, metastatic malignant glial tumors, multifocal gliomas and bithalamic gliomas are eligible for the study. Diffuse midline gliomas with H3K27M mutation are not eligible. Anaplastic ganglioglioma and anaplastic pleomorphic astrocytoma will be eligible.
7. Local histological diagnosis after either stereotactic biopsy or surgical procedure has been confirmed centrally by a designated reference pathologist.
8. Able to commence trial treatment within 6 weeks following the last major surgery.
9. Adequate Bone Marrow Function : Hemoglobin >/= 10 g/dL (transfusion independent), Neutrophil count >/= 1.0 x 10^9/L.

   Platelet count >/= 1.0 x 10^9/L (transfusion independent)
10. Absence of Coagulation Disorder
11. Adequate Liver Function : AST </= 2.5x institutional ULN for age, ALT </= 2.5x institutional ULN for age, Total Bilirubin </= 1.5x institutional ULN for age
12. Adequate Renal Function : Serum creatinine must be </= 1.5x ULN for age, absence of clinically significant proteinuria as defined by a screening early morning urine (first sample) dipstick urinalysis of </= 2

Exclusion Criteria:

1. Any disease or condition that contraindicates the use of the study medication/treatment (for TMZ, see the approved product labelling) or places the patient at an unacceptable risk of experiencing treatment related complications.
2. Patients should not be on high-dose steroids (ie > 1mg/kg) before study entry; doses should be stable for at least two weeks or decreasing.
3. Low probability of protocol compliance.
4. Radiological evidence of surgically related intracranial bleeding (excluding asymptomatic, resolving hemorrhagic changes associated with recent surgery and the presence of punctuate hemorrhage in the tumor).
5. Subjects with concommitant second malignancies are excluded unless a complete remission is achieved as it is empirically determined based on the malignancy and treatment provided prior to study entry and no additional therapy is required or anticipated to be required during the study period.
6. Previous cranial irradiation.
7. Any known auto-immune disease, previous or ongoing.
8. Known chronic inflammatory digestive disease, previous or ongoing.
9. Chronic asthma receiving corticotherapy, even only with inhalation.
10. Vaccinated with live attenuated vaccines within 4 weeks of the first dose of study drug
11. Pregnant or breastfeeding women
12. Known hypersensitivity to any component of the products (study drug or ingredients)
13. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening).
14. Patients who are currently receiving another investigational drug or anticancer agent
15. Patient who have an uncontrolled infection
16. Patient with known human immunodeficiency virus (HIV) / AIDS infection or acute / chronic Hepatitis B or C

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | The clinical activity of the combined treatment will be evaluated by the 1-year event free survival (EFS)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Gustave Roussy, Villejuif, Val De Marne
  - CHU Angers, Angers
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - CHU Hautepierre, Strasbourg
  - Hôpital des enfants, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided